CLINICAL TRIAL: NCT07086976
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study With an Open-label Period and Long-term Extension to Assess the Efficacy and Safety of Rilzabrutinib in Participants With Warm Autoimmune Hemolytic Anemia (wAIHA)
Brief Title: A Study to Investigate the Efficacy, Safety, and Pharmacokinetics of Oral Rilzabrutinib Compared With Placebo in Participants 18 Years of Age and Older With Warm Autoimmune Hemolytic Anemia
Acronym: LUMINA 3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17360; U1111-1314-5112 (Registry Identifier: ICTRP); 2024-517972-39 (Registry Identifier: CTIS)
Record Dates: First submitted 2025-07-17; First posted 2025-07-25 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Haemolytic Anaemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- rilzabrutinib (Experimental): Oral rilzabrutinib BID
  Interventions: Drug: rilzabrutinib
- placebo (Placebo Comparator): Oral placebo BID
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rilzabrutinib — Pharmaceutical form:tablet-Route of administration:oral
  Other Names: SAR444671
  Arms: rilzabrutinib
Drug: placebo — Pharmaceutical form:tablet-Route of administration:oral
  Arms: placebo

SUMMARY:
This is a parallel-group, Phase 3, double-blind, 2-arm study to investigate the efficacy, safety, PK and PD of oral rilzabrutinib in achieving durable Hb response (DHR) compared with placebo in approximately 90 male and female participants ≥ 18 years of age with a confirmed diagnosis of primary wAIHA.

Following a 4-week screening period, eligible participants will be randomized in a 2:1 ratio to receive rilzabrutinib or placebo in primary analysis period (PAP) for a duration of up to 24 weeks. All participants who completed PAP will then continue in open-label period (OLP) to receive rilzabrutinib for a duration of 28 weeks. Upon the completion of OLP, only participants who demonstrate Hb increase during the last 8 weeks of OLP per specified criteria in the protocol will be eligible to continue in long-term extension (LTE) of the study. The duration of the LTE period will be from the first-participant-in (FPI)-LTE until the last participant completes 52 weeks in LTE. The safety follow-up period of this study following treatment completion or discontinuation will be 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants with a documented (confirmed) diagnosis of primary wAIHA for at least 3 months.
* Participants who have previously failed to maintain a sustained response after treatment with CS (CS-resistance [defined as failure to obtain hemoglobin response within 3 weeks on at least 1 mg/kg or 60 mg prednisone or equivalent per day], CS-dependent wAIHA [defined as need to continue on prednisone or equivalent at a dose of >10 mg/day to maintain a response]), or are intolerant or ineligible to CS (defined as with contraindications, pre-existing medical conditions or CS-related complications that may render CS intolerant or ineligible per the best clinical judgement of the investigators).
* Participants with Eastern Cooperative Oncology Group (ECOG) performance status Grade 2 or lower.
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Participants with clinically significant medical history or ongoing chronic illness that would jeopardize the safety of the participant or compromise the quality of the data derived from his or her participation in the study as determined by the Investigator.
* Participants with medical history of lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for the past 3 years.
* Participants with symptomatic herpes zoster within 3 months prior to screening.
* Participants with secondary wAIHA from any cause including drugs, Evans Syndrome, lymphoproliferative disorders (low count monoclonal B-cell lymphocytosis is allowed), infectious or autoimmune disease, or active hematologic malignancies. Participants with positive antinuclear antibodies but without a definitive diagnosis of an autoimmune disease are allowed.
* Participants with history of myelodysplastic syndrome.
* Participants with uncontrolled or active HBV infection or Active HCV infection.
* HIV infection.
* Participants with history of solid organ transplant.
* Participants with a history of active or latent tuberculosis (TB).
* Concurrent treatment with other experimental/investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to treatment start. Participants who previously received treatment with BTK inhibitors for wAIHA before Day 1 (randomization) are not eligible.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-08-18 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-12-26 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving DHR. DHR is defined as an increase of Hb by ≥2 g/dL from baseline on at least two thirds of evaluable scheduled visits between Week 12 and Week 24 (inclusive) in the PAP | By Week 24
  DHR is defined as an increase of Hb by ≥2 g/dL from baseline on at least two thirds of evaluable scheduled visits between Week 12 and Week 24 (inclusive) in the PAP in the absence of rescue medication and transfusion.

SECONDARY OUTCOMES:
Proportion of participants achieving overall Hb response (response [R] or complete response [CR]) by Week 24 of treatment in the PAP | By Week 24
  Response is defined as an increase in Hb by ≥2 g/dL from baseline in the absence of transfusion and rescue medication.
  Complete Response is defined as Hb ≥12 g/dL (women) or ≥13 g/dL (men) without evidence of hemolysis (ie, normal indirect bilirubin, lactate dehydrogenase [LDH], haptoglobin, and reticulocytes), in the absence of transfusion and rescue medication.
The time taken (days) to achieve the first Hb increase by ≥2 g/dL from baseline during the PAP in the previous 14 days and in the absence of rescue medication in the previous 6 weeks | Until Week 24
Change from baseline in fatigue total score as measured by Functional Assessment of Chronic Illness Therapy (FACIT) - fatigue at Week 24 | Baseline to Week 24
Change from baseline in levels of LDH at Week 24 | Baseline to Week 24
Proportion of participants requiring use of rescue therapy after Week 4 of treatment during the PAP | Until Week 24
Change from baseline in dyspnea severity score as measured by FACIT-Dyspnea at Week 24 | Baseline to Week 24
Incidence of treatment-emergent adverse events (TEAE), treatment-emergent serious adverse events (SAEs), treatment-emergent adverse events of special interest, as well as clinical laboratory evaluations, vital sign, physical exam, and electrocardiograms | Until Week 104

CONTACTS AND LOCATIONS:
Locations (78):
- United States (15):
  - Mayo Clinic- Site Number : 8400032, Phoenix, Arizona
  - Noble Clinical Research- Site Number : 8400003, Tucson, Arizona
  - City of Hope- Site Number : 8400023, Duarte, California
  - University of Southern California (USC)- Site Number : 8400007, Los Angeles, California
  - The Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center- Site Number : 8400006, Torrance, California
  - Yale University School of Medicine- Site Number : 8400027, New Haven, Connecticut
  - Bioresearch Partners- Site Number : 8400009, Hialeah, Florida
  - Oncology and Hematology Associates of West Broward, PA- Site Number : 8400005, Tamarac, Florida
  - University of Michigan- Site Number : 8400014, Ann Arbor, Michigan
  - Mayo Clinic- Site Number : 8400008, Rochester, Minnesota
  - Montefiore Medical Center- Site Number : 8400011, The Bronx, New York
  - Ohio State University Hospital East- Site Number : 8400020, Columbus, Ohio
  - Baptist Memorial Hospital- Site Number : 8400018, Memphis, Tennessee
  - University of Texas Health Science Center at San Antonio- Site Number : 8400015, San Antonio, Texas
  - Gundersen Health System- Site Number : 8400033, La Crosse, Wisconsin
- Argentina (3):
  - Investigational Site Number : 0320002, CABA, Buenos Aires F.D.
  - Investigational Site Number : 0320003, Ciudad Autonoma Buenos Aires, Buenos Aires F.D.
  - Investigational Site Number : 0320001, Rosario, Santa Fe Province
- Austria (2):
  - Investigational Site Number : 0400001, Vienna
  - Investigational Site Number : 0400002, Vienna
- Brazil (3):
  - Centro Estadual de Hemoterapia e Hematologia Marcos Daniel Santos - HEMOES- Site Number : 0760002, Vitória, Espírito Santo
  - HC UFG - Hospital Das Clinicas de Goias- Site Number : 0760001, Goiânia, Goiás
  - Hospital das Clinicas de Sao Paulo- Site Number : 0760003, São Paulo, São Paulo
- China (12):
  - Investigational Site Number : 1560001, Beijing
  - Investigational Site Number : 1560007, Chengde
  - Investigational Site Number : 1560005, Guangzhou
  - Investigational Site Number : 1560011, Guangzhou
  - Investigational Site Number : 1560009, Hohhot
  - Investigational Site Number : 1560003, Nanchang
  - Investigational Site Number : 1560012, Nanchang
  - Investigational Site Number : 1560004, Suzhou
  - Investigational Site Number : 1560002, Tianjin
  - Investigational Site Number : 1560010, Wuhan
  - Investigational Site Number : 1560006, Xi'an
  - Investigational Site Number : 1560008, Zhengzhou
- Czechia (2):
  - Investigational Site Number : 2030002, Prague, Cardiff [Caerdydd Gb-crd]
  - Investigational Site Number : 2030001, Brno
- Denmark (3):
  - Investigational Site Number : 2080003, Aarhus N
  - Investigational Site Number : 2080002, Copenhagen
  - Investigational Site Number : 2080001, Odense C
- Germany (2):
  - Investigational Site Number : 2760003, Charlottenburg
  - Investigational Site Number : 2760001, Essen
- Greece (5):
  - Investigational Site Number : 3000002, Athens
  - Investigational Site Number : 3000005, Larissa
  - Investigational Site Number : 3000004, Pátrai
  - Investigational Site Number : 3000003, Pátrai
  - Investigational Site Number : 3000001, Thessaloniki
- Investigational Site Number : 3480002, Debrecen, Hungary
- Israel (4):
  - Investigational Site Number : 3760001, Afula
  - Investigational Site Number : 3760007, Haifa
  - Investigational Site Number : 3760005, Kfar Saba
  - Investigational Site Number : 3760002, Tel Aviv
- Italy (8):
  - Investigational Site Number : 3800002, Meldola, Forlì-Cesena
  - Investigational Site Number : 3800004, Florence, Tuscany
  - Investigational Site Number : 3800010, Genova
  - Investigational Site Number : 3800001, Milan
  - Investigational Site Number : 3800005, Napoli
  - Investigational Site Number : 3800009, Novara
  - Investigational Site Number : 3800007, Trieste
  - Investigational Site Number : 3800003, Vicenza
- Japan (8):
  - Investigational Site Number : 3920002, Fukushima, Fukushima
  - Investigational Site Number : 3920006, Kanazawa, Ishikawa-ken
  - Investigational Site Number : 3920008, Okayama, Okayama-ken
  - Investigational Site Number : 3920003, Suita-shi, Osaka
  - Investigational Site Number : 3920001, Iruma-gun, Saitama
  - Investigational Site Number : 3920005, Yamagata, Yamagata
  - Investigational Site Number : 3920010, Kofu, Yamanashi
  - Investigational Site Number : 3920015, Fukuoka
- Netherlands (2):
  - Investigational Site Number : 5280002, Amsterdam
  - Investigational Site Number : 5280003, Leiden
- Investigational Site Number : 6160005, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland
- Spain (5):
  - Investigational Site Number : 7240001, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240005, Barakaldo, Bizkaia
  - Investigational Site Number : 7240007, Majadahonda, Madrid
  - Investigational Site Number : 7240004, Madrid / Madrid, Madrid, Comunidad de
  - Investigational Site Number : 7240003, Seville
- Sweden (2):
  - Investigational Site Number : 7520003, Malmo
  - Investigational Site Number : 7520001, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Warm Autoimmune Hemolytic Anemia Website — https://www.sanofistudies.com/OEA7/
- See also: EFC17360 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26781&tenant=MT_SNY_9011